CLINICAL TRIAL: NCT03583437
Title: The Effect of Physical Activity on the Liver and the Heart's Metabolism of Fatty Acids in Obese With and Without NAFLD
Brief Title: Hepatic and Cardiac Metabolic Flexibility in Obese With NAFLD.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: jeyanrk
Record Dates: First submitted 2018-05-22; First posted 2018-07-11 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: NAFLD - Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Experimental: 1 Healthy male volunteers Behavioral: Exercise Moderate Intensity Exercise (50 % af VO2max) for 90 minutes before and after PET scanning, Experimental: 2 Healthy female volunteers Moderate Intensity Exercise (50 % af VO2max) for 90 minutes before and after a PET scanning.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy male volunteers (Experimental): Behavioral: Exercise Moderate Intensity Exercise (50 % af VO2max) for 90 minutes before and after PET scanning.
  Interventions: Behavioral: Exercise
- Healthy female volunteers (Experimental): Behavioral: Exercise Moderate Intensity Exercise (50 % af VO2max) for 90 minutes before and after PET scanning.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Moderate Intensity Exercise (50 % af VO2max) for 90 minutes

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) covers a spectrum from reversible hepatic steatosis to inflammation and fibrosis termed steatohepatitis (NASH) and cirrhosis. New evidence indicates that NAFLD is associated with development of heart failure, abnormal ventricular glucose and fatty acid (FA) utilisation and cardiosteatosis. The mechanisms behind cardiac involvement and the progression from NAFLD to NASH are poorly understood but must include altered cardiac and intrahepatic lipid handling. In collaboration with renowned research groups from Oxford, Mayo Clinic and Copenhagen investigators plan comprehensive kinetic studies of heart and liver FA uptake and oxidation, ventricular function and substrate utilisation, and hepatic triglyceride (TG) secretion in order to assess mechanisms governing cardiac and hepatic lipid and glucose trafficking in subjects with NAFLD and NASH and the relationship with heart function. In addition, the investigators will assess skeletal muscle and adipose tissue enzyme activities, gene expression and protein concentrations in these subjects to define mechanisms involved in the cross-talk between heart, liver, muscle and adipose tissues. Investigators will address these questions using innovative tracer techniques (11Cpalmitate, 11C acetate, 18FDG glucose PET tracers and TG tracers) in combination with hepatic vein catherisation to study cardiac and liver substrate trafficking, as well as NMR spectroscopy, echocardiography, muscle and fat biopsies in combination with state-of-the art muscle and adipose tissue enzyme kinetics, gene- and protein expression. Effects of acute exercise will be assessed. The overarching goals are to define abnormalities and differences between NAFLD and NASH in hepatic lipid (FA and TG) metabolism and to assess the effect of exercise on both hepatic, cardiac and adipose and skeletal muscle lipid and substrate utilisation.

ELIGIBILITY:
Inclusion Criteria:

* 10 obese subject men/women with NAFLD (MR spectroskopi, fibro scanner) (BMI > 30).
* 10 obese subject men/women without NAFLD (MR spectroskopi, fibro scanner) (BMI > 30).
* age between 40-70 years
* Written consent before the start of the study

Exclusion Criteria:

* known current disease
* Fixed Medical drug consumption, statins and antihypertensive drugs (non-beta blocker). However, pause 3 weeks before the examination date
* Blood donation within the last 3 months prior to the study
* Participation in experiments involving radioactive isotopes within the last 6 months
* Alcohol abuse (over 21 items per week for men and 14 for women)
* Smoking
* Weight over 130 kg
* Cancer patients
* Large intake of medication

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2020-09-07 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
The effect of physical activity on the heart's metabolism of fatty acids in obese with and without NAFLD | 2 years
  Primary outcome:
  - Fatty acid uptake (mg/kg/min) in the Heart in obese with and without NAFLD

SECONDARY OUTCOMES:
To determine the effect of an acute exercise bout on the improvement of cardiac FA utilization in obese with and without NAFLD. | 2 years
  Fatty acid oxidation (µmol/min) in the Heart in obese with and without NAFLD.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Diabetes and Hormone diseases in Aarhus University Hopital, Skejby, Aarhus N, Denmark